CLINICAL TRIAL: NCT00135785
Title: A Randomized, Double-Blind, Placebo-Controlled Evaluation of Bupropion vs Placebo for the Treatment of Methamphetamine Dependence
Brief Title: Effectiveness of Bupropion Combined With Behavioral Therapy for Treating Methamphetamine Dependence - 2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Collaborators: University of California, Los Angeles (Other)
Responsible Party: Dr Steven Shoptaw, UCLA Department of Family Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NIDA-18185-2; P50-DA018185-2; DPMC; P50DA018185 (NIH)
Record Dates: First submitted 2005-08-23; First posted 2005-08-26 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2009-09

CONDITIONS: Methamphetamine
MeSH Terms: interventions — Bupropion

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Bupropion
  Interventions: Drug: Bupropion
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Bupropion
  Arms: 1
Drug: Placebo
  Arms: 2

SUMMARY:
Methamphetamine is an addictive stimulant drug that strongly activates certain parts of the brain. The purpose of this study is to determine the effectiveness of bupropion in combination with behavioral therapy for the treatment of methamphetamine addiction.

DETAILED DESCRIPTION:
Methamphetamine is a drug that causes excess amounts of the neurotransmitters dopamine and norepinephrine to be released into the brain. This overload produces unusual alertness and feelings of elation. When the body undergoes methamphetamine withdrawal, it experiences a reduction in dopamine and norepinephrine. Bupropion is an antidepressant used for the treatment of depression and smoking cessation. Because it functions by increasing the release of dopamine and norepinephrine in the brain, bupropion is likely to decrease the negative effects of methamphetamine withdrawal. The purpose of this study is to evaluate the efficacy of bupropion combined with contingency management (CM) and cognitive behavioral counseling (CBT) as a means of treating methamphetamine dependence.

An initial 2-week screening process will involve participants providing urine samples and completing physical and psychological assessments. If deemed eligible for the remainder of this double-blind study, participants will be randomly assigned to receive either bupropion or placebo over the course of 12 weeks. Participants in both the bupropion and placebo groups will receive contingency management and cognitive behavioral counseling. Participants will report to one of two clinical research sites three times per week. At each visit, participants will be examined by the study staff, provide a urine sample, and receive individual cognitive behavioral counseling sessions. At the end of 12 weeks, treatment will be stopped. Participants will return to the study site 30 days later for evaluation and to be assessed for any possible lingering side effects.

ELIGIBILITY:
Inclusion Criteria:

* Meets DSM-IV criteria for methamphetamine dependence
* Females must use an effective method of contraception

Exclusion Criteria:

* History of or current medical condition that might interfere with safe participation, such as active tuberculosis, unstable heart or liver disease, unstable diabetes, symptomatic AIDS (non-symptomatic HIV infection is not an exclusion), or greater than 8 times the upper limit of normal in liver screening function tests (SGOT or SGPT)
* Current neurological disorder (e.g., organic brain disease, dementia)
* Major psychiatric disorder unrelated to substance abuse, such as schizophrenia or bipolar disorder (assessed by the SCID and a medical history)
* Suicide attempt within the month prior to enrollment and/or currently suicidal (assessed by the SCID and the BDI II)
* Currently on prescription medication that might interact with the study drug
* Currently dependent on cocaine, opiates, alcohol, or benzodiazepines, as defined by DSM-IV-TR criteria
* History of alcohol dependence within past three years
* History of seizure disorders
* History of anorexia or bulimia
* Current hypertension uncontrolled by medication
* History of sensitivity to bupropion
* Pregnant or breastfeeding

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2005-10; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Addiction severity, Week 16
Drug use, Week 16

CONTACTS AND LOCATIONS:
Overall Officials: Steve Shoptaw, Ph.D., Principal Investigator — University of California, Los Angeles
Locations (2):
- United States (2):
  - UCLA Medical Center, Los Angeles, California
  - Rancho Cucamonga Clinic, Rancho Cucamonga, California